CLINICAL TRIAL: NCT05100121
Title: To Live Better After Prostate Cancer Treatment: a Randomized Pilot Trial of Supportive and Person-centered Care Intervention in Primary Care
Brief Title: To Live Better After Prostate Cancer Treatment:
Acronym: CAPPRIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Ann Langius-Eklöf, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Dnr-2019-0037
Record Dates: First submitted 2021-10-08; First posted 2021-10-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Prostate Cancer
Keywords: mobile health; Prostate cancer; Symptom management; primary care; self- management; Support
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention consists of standard care and an app for routine symptom reporting, weekly the first month and thereafter as mutually agreed, at minimum once a month in one year, with instant self-managment advice in combination with supportive care with a study-specific nurse. At health dialogues with the nurse, the patient-reported assessments in the app will be used to discuss the individual's current situation and to plan eventual additional actions needed. The intervention will last for 6 months.
  Interventions: Device: Interactive app; Other: Supportive Care
- Control (No Intervention): The participants in the control group will only receive standard care. Usually after ended curative treatment the follow-up is a blood sample (PSA) every three or six months the first year, this can be handled either by a nurse or a physician in secondary care. Most hospitals also have one physical meeting with a physician three months after ended treatment (Regional Cancer Centers, 2020). All patients are allocated a contact nurse with a telephone number to contact when needed.

INTERVENTIONS:
Device: Interactive app — In the app, the patients will report frequency and distress on commons concerns regarding urine dysfunction, bowel dysfunction, emotional distress, sleep, pain, loss of appetite, hot flashes/sweating, edema, and sexual dysfunction. Free text comments will also be possible to make to cover the patients' other potential needs. Questions regarding symptoms of acute character that might need to be treated quickly like severe pain, blood in stool and urine, and involuntary weight loss will also be asked for to timely detect and treat signs of for example cancer relapse. Information about the concerns will be included in the app containing; a) general information of why they have the side effect and what it means b) evidence-based advice about self-management; c) when they should contact health care providers, and d) further information linked to reliable documents and web pages.
  Arms: Intervention
Other: Supportive Care — During the health dialogues with the nurse, the patient reported assessments will be used to discuss the individual's current situation and to plan eventual additional actions needed such as support from a physiotherapist, social worker, dietitian or if a visit to the physician if needed. This is documented in the patients health record.
  Arms: Intervention

SUMMARY:
It is evident that patients receiving treatment for cancer have symptoms that often are undetected. Furthermore, many survivors from cancer have ongoing poor health and well-being and long-term rehabilitation and support should not be neglected to prevent recurrence and increase survival. There are good reasons to believe that routine collection of relevant patient-reported symptoms facilitates person-centered care where the patient is a participatory member of the team. This study aims to pilot-test a supportive intervention in primary care for six months during the first year after primary treatment for prostate cancer in primary care and compare it to standard care only. The intervention consists of symptom reporting and self-management in an app in combination with health dialogues with a study-specific nurse at a primary care centre.

DETAILED DESCRIPTION:
Prostate cancer is the most common form of cancer in Sweden and the most common form of cancer among men in Sweden, representing approximately 30 percent of all cancer cases among men. The median age for being diagnosed with prostate cancer is around 69. The treatments available for prostate cancer can impact the patients; quality of life (QoL) (Katz, 2007). After surgery and radiation treatment, the function of the bowel and bladder is affected. Erectile dysfunction is common after surgery, radiation, and hormonal therapy. Symptoms and side effects can start quite suddenly, get improved, but also persist a long time after treatment.

Psychosocial support to patients during the treatment shows different results, some with positive effects on QoL by psychoeducational or nurse-delivered interventions and some with no effect at all.

Patient-reported outcome (PRO) is an outcome that is reported by the patients. Previous research on collecting PROs through an interactive application during treatment for breast cancer, pancreatic cancer, and prostate cancer shows promising results such as reduced symptom burden and improved QoL as well as on survival. A synthesis of current research on web-based interventions shows how important it is that content is specific to the patients' needs and delivered at the right stage in the cancer trajectory and emphasize user involvement in the developmental phase.

The aim is to pilot-test routine assessment of patient reported symptoms and support in self-management assisted by digital technology for six months during the first year after primary treatment for prostate cancer in combination with helath dialouges with a study-specific nurse at the primary care centre.

The primary objective is to evaluate the acceptability and feasibility of digital and nurse-led support intervention in primary care during the first after primary treatment. The secondary objectives of these trials are to (i) evaluate the potential efficacy of the intervention and (ii) obtain estimates for secondary outcome measures and potential mediators and moderators to be used in a future trial and (iii) evaluate the feasibility of such assessments.

There are around 250 Primary Health Care Centers (PHCC) in Stockholm and to achieve representative PHCCs for randomization a Care Need Index (CNI) is used. CNI is a model that measures healthcare needs for the distribution of primary care resources to the population with the biggest need. High CNI index equals low socioeconomic status and low CNI index equals high socioeconomic status. The study has a prospective, cluster randomized controlled pilot trial design The studies have two parallel arms; the intervention plus standard care (intervention group); and standard care alone (control group). Approximately ten PHCCs will be matched on CNI index and the number of patients allocated to the PHCCs.

ELIGIBILITY:
Inclusion Criteria:

* patients with prostate cancer at the end of curative treatment
* able to read and understand Swedish
* considered being physically, psychologically and cognitively able to participate in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study is about men with prostate cancer.
Enrollment: 40 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Acceptability E -scale | 6 months
  The Acceptability e-scale is a questionnaire with 6 items that evaluate the acceptability of a system. Items are scored using a Likert scale ranging from 1-5 with higher values indicating higher acceptability.
System Usability Scale (Q5 and Q10) | 6 months
  The System Usability Scala is a questionnaire with ten item that evaluate the usability of a system. Items are scored using a Likert scale ranging from 1-5. Only question 5 and 10 will be included in this study.
Interviews | 7 months
  To assess acceptability and feasibility, the participants in the intervention group and the study specific nurses will be interviewed about their experinece using the Interaktor system and about the health dialouges.
Other feasibility measures | Through study completion, an avrage of 24 months
  To evaluate the feasibility of the future trial methodology, enrollment, recruitment, and withdrawal rates will be documented. Other feasibility measures include completion rates and missing data in each study questionnaire. Objective measures will be extracted from the logged data in the app, i.e., the number of reports sent (adherence), self-managment advice viewings, and notes from the study-specific nurses.

SECONDARY OUTCOMES:
Symptom burden measured by the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire - Prostate Module | Baseline, 3 months, 6 months, 12 months, 18 months, and 24 months
  The questionnaire has 25 items and evaluates specific prostate cancer symptoms related to treatment such as sexual function and bladder and bowel problem. Items are scored using a Likert scale ranging from 1-4 with higher values indicating more burden of symptoms and divided in six sub-scales.
Quality of Life measured by the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire | Baseline, 3 months, 6 months, 12 months, 18 months, and 24 months
  The questionnaire has 30 items divided in five functional scales (physical, role, emotional, social, and cognitive), eight symptom scales (fatigue, nausea and vomiting, pain, insomnia, appetite loss, constipation, diarrhea), financial impact of the disease, and a global health status/QoL scale. Questions are scored using a Likert scale ranging from 1-4 with higher values indicating lower QoL.
The Patient Activation Measure (PAM -13) | Baseline, 3 months, 6 months, 12 months, 18 months, and 24 months
  The PAM-13 questionnaires has 13 items measure knowledge, skils, beliefs, and confidence in managin health and healthcare.
Quality of life measured measured by the EuroQol 5-Dimension Questionnaire (EQ-5D-5L) | Baseline, 3 months, 6 months, 12 months, 18 months, and 24 months
  For this study used together with direct costs to analyse Quality of adjusted life years by weighting life expectancy of a patient against estimation of a persons' health related Quality of Life score.
The Sence of Coherence Scale (SOC-13) | Baseline, 3 months, 6 months, 12 months, 18 months, and 24 months
  The SOC-13 questionnaire measure overall coping ability.
Health Literacy CCHL (5-items) | Baseline, 3 months, 6 months, 12 months, 18 months, and 24 months
  The questionnaire has five items measuring the ability to read and understand information regarding health, disease and health care

CONTACTS AND LOCATIONS:
Overall Officials: Ann Langius-Eklöf, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Health Care Services Stockholm County (SLSO), Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Langius-Eklof A, Craftman AG, Gellerstedt L, Kelmendi N, Rooth K, Gustavell T, Sundberg K. Digital and nurse-led support intervention in primary care during the first year after curative intent treatment for breast or prostate cancer: study protocol of two cluster randomised controlled pilot trials. BMJ Open. 2025 Feb 22;15(2):e090848. doi: 10.1136/bmjopen-2024-090848. PMID 39986997